CLINICAL TRIAL: NCT02355795
Title: Diets With a Spectrum of Fat Intake for Preventing Obesity: A Randomized Controlled-feeding Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Collaborators: National Basic Research Program, China (Other); National Natural Science Foundation of China (Other Government); Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Duo li, Professor, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: DUOLI201501
Record Dates: First submitted 2015-01-25; First posted 2015-02-04 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: weight change; diet; dietary fat; feeding design
MeSH Terms: conditions — Body Weight Changes | interventions — Diet, Fat-Restricted; Diet, High-Fat

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (3):
- low-fat diet (Experimental): Participants will be provided low-fat diet for 6 months
  Interventions: Behavioral: low-fat diet
- moderate-fat diet (Experimental): Participants will be provided moderate-fat diet for 6 months
  Interventions: Behavioral: moderate-fat diet
- high-fat diet (Experimental): Participants will be provided high-fat diet for 6 months
  Interventions: Behavioral: high-fat diet

INTERVENTIONS:
Behavioral: low-fat diet — Energy from total fat, protein and carbohydrates are 20%, 14% and 66%, respectively
  Arms: low-fat diet
Behavioral: moderate-fat diet — Energy from total fat, protein and carbohydrates are 30%, 14% and 56%, respectively
  Arms: moderate-fat diet
Behavioral: high-fat diet — Energy from total fat, protein and carbohydrates are 40%, 14% and 46%, respectively
  Arms: high-fat diet

SUMMARY:
The aim of the current study is to evaluate the effects of diets with three levels of dietary fat on weight change and related cardiometabolic risk factors in a 6-month randomized controlled-feeding trial.

ELIGIBILITY:
Inclusion criteria:

* Students in Zhejiang University or working stuff in the Chinese PLA General Hospital
* 18 ≤ age ≤ 35
* Body Mass Index < 28*
* Are willing to eat all of the study foods even when full
* Are willing to eat only foods provided
* Are willing to avoid strenuous activity during the 6-mo intervention Exclusion criteria：
* Systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg
* Total cholesterol ≥ 239 mg/dL
* Low-density lipoprotein cholesterol ≥ 159 mg/dL
* Triglycerides ≥ 199 mg/dL
* Blood glucose ≥ 110 mg/dL
* Change in body weight exceeding ± 10% during the prior year
* Energy intake is too low or too high
* Unwillingness or special requirement for diet that could not be modified
* Poor adherence during the recruiting meeting or unsatisfactory completion of keeping food diary or filling questionnaire at any time before randomization
* Eating disorder or any psychosocial or scheduling factors that could impede study outcomes
* Have a history of diagnosed CVD, diabetes, cancer or inflammatory diseases
* Have a history of a mental illness
* Have diagnosed endocrine, pulmonary or hematological disease
* Have diagnosed bowel disease or malabsorption that would prevent the participants from complying with the dietary restrictions of the feeding trial
* Renal or liver insufficiency
* Other chronic disease thought to interfere with the effect of the diet or with participation or adherence
* Current use of supplements or anti-inflammation medications or medications affecting glucose, lipid metabolism and blood pressure
* Smoking or alcoholic beverage intake >1 times per week
* Current or planned pregnancy prior to end of study, or breast-feeding
* Irregular menstrual cycles
* Have birth control medication

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 307 (Actual)
Dates: Start 2014-11; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
body weight in kilograms as measured by a calibrated scale | 0,1,2,3,4,5,and 6 months
  change from baseline will be reported

SECONDARY OUTCOMES:
waist circumference as measured by an anthropometric measuring tape | 0,1,2,3,4,5,and 6 months
  change from baseline will be reported
blood pressure as measured by a validated automated sphygmomanometer | 0,1,2,3,4,5,and 6 months
  change from baseline will be reported
fasting blood lipids as measured by a clinical chemistry analyzer | 0,1,2,3,4,5,and 6 months
  change from baseline will be reported
fasting glucose, insulin, glycated serum protein as measured by an immunology analyzer | 0,1,2,3,4,5,and 6 months
  change from baseline will be reported
adiponectin, leptin as measured by ELISA kits | 0,1,2,3,4,5,and 6 months
  change from baseline will be reported

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang University, Hangzhou, Zhejiang, China

REFERENCES:
- [Derived] Wan Y, Yuan J, Li J, Li H, Zhang J, Tang J, Ni Y, Huang T, Wang F, Zhao F, Li D. Unconjugated and secondary bile acid profiles in response to higher-fat, lower-carbohydrate diet and associated with related gut microbiota: A 6-month randomized controlled-feeding trial. Clin Nutr. 2020 Feb;39(2):395-404. doi: 10.1016/j.clnu.2019.02.037. Epub 2019 Feb 27. PMID 30876827
- [Derived] Wan Y, Wang F, Yuan J, Li J, Jiang D, Zhang J, Li H, Wang R, Tang J, Huang T, Zheng J, Sinclair AJ, Mann J, Li D. Effects of dietary fat on gut microbiota and faecal metabolites, and their relationship with cardiometabolic risk factors: a 6-month randomised controlled-feeding trial. Gut. 2019 Aug;68(8):1417-1429. doi: 10.1136/gutjnl-2018-317609. Epub 2019 Feb 19. PMID 30782617
- [Derived] Wan Y, Wang F, Yuan J, Li J, Jiang D, Zhang J, Huang T, Zheng J, Mann J, Li D. Effects of Macronutrient Distribution on Weight and Related Cardiometabolic Profile in Healthy Non-Obese Chinese: A 6-month, Randomized Controlled-Feeding Trial. EBioMedicine. 2017 Aug;22:200-207. doi: 10.1016/j.ebiom.2017.06.017. Epub 2017 Jun 20. PMID 28655596